CLINICAL TRIAL: NCT00728871
Title: The Correlations Between HPV L1-Specific Immunologic Responses in Cervical Cancer and CIN Patients and Their Prognosis
Brief Title: The Correlations Between HPV L1-Specific Immunologic Responses in Cervical Cancer and Cervical Intraepithelial Neoplasia (CIN) Patients and Their Prognosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Chi-An Chen/Professor, National Taiwan Unviersity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9461700838
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Cervical Cancer; Cervical Intraepithelial Neoplasia
Keywords: cervical cancer, HPV, immunity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia; Papillomavirus Infections

INTERVENTIONS:
Procedure: peripheral blood isolation — To isolate serum from patient peripheral blood to test the titer of HPV infection and cytokine expression

SUMMARY:
A. To investigate the relationship between serum titer of anti-HPV16 antibody and clinicopathological factors of cervical cancer patients.

B. To investigate that if the serum titer of anti-HPV16 antibody could be a prognostic factor in the cervical cancer patients.

C. To investigate the serum titer of anti-HPV16 antibody in HPV16-infected populations with various disease status such as infection only, precancerous lesion, and early and advanced cervical cancer.

DETAILED DESCRIPTION:
Cervical cancer is the most frequent neoplasm of the women in Taiwan and in the world. Cervical cancer affects half a million women each year and results in about 200,000 worldwide and it also influences about 2,700 women and about 1,000 women dying of cervical cancer each year and in Taiwan. There is strong evidence suggesting that this cancer is 100% attributable to infection with certain types of human papillomavirus (HPV); in fact, the World Health Organization (WHO) has very recently recognized that this cancer is caused by HPV. There are around 100 different HPV-types, of which around 40 types infecting the anogenital tract and causing cervical lesions and cervical cancer have been called High Risk HPV (i.e., HR-HPV-16, -18, -31, -33, and -58). From recent years, there is compelling evidence that infection with human papillomavirus (HPV) is a major etiologic factor in the development of cervical intraepithelial neoplasia (CIN) and cervical carcinoma.

As in most virus induced diseases, an adequate immune response is likely to play a key role in clearance of HPV infections and HPV-related lesions. This assumption is born out by both epidemiological studies and animal models. Immune compromised patients such as HIV infected women, organ transplant recipients, and patients suffering other forms of malignancies, are at higher risk of developing CIN lesions and invasive cervical cancer. Moreover, several studies establish the existence of natural HPV-specific immunity in humans. Immune responses of the host are indeed critical in the virus-related infectious diseases. The immune response against HPV antigens is Human leukocyte antigen restricted. Consequently, the HLA class I and II phenotype may be correlated with an effective immune response against HPV associated cervical lesions. Differences in the recognition of foreign antigen, such as those contributed by alleles at the HLA class I or II loci, might be proposed to affect the risk of developing cervical cancer. Studies by different groups on associations between certain HLA alleles and susceptibility to, or protection against CIN lesions and cervical carcinoma, reveal varying conclusions and warrant further research.

Most potentially oncogenic, persistent, long-term HPV infections induce an antibody response against virus proteins which can be detected by ELISA test and can be a good indicator of past as well as current infections and chronic active infection, associated with the presence of cervical lesions and the high risk of acquiring cervical cancer. In fact, it has been reported that women who are seropositive for HPV-16 present a higher risk of developing cervical carcinoma than seronegative women. L1-viral capsid proteins are one of the targets for antibodies induced by persistent HPV genital infection.

The L1 protein represents more than 90% of the total protein on the surface of the virus. This protein is able to assemble itself, forming virus-like particles (VLPs). VLPs, mainly type 16, have been broadly used for studying the antibody response induced by genital HPVinfection. The VLP-antibody presence is stable in time, correlated with the number of sexual partners, and associated with persistent infection, viral load, and development of neoplasic lesions; this is rarely found in patients suffering from transitory infections. Seropositivity occurs more frequently in patients who have progressed to CIN III and invasive cancer than in those suffering from CIN I or CIN II and the antibody response is significantly higher in women having a higher viral load than those with lower viral load. Prospective studies have shown that 70-90% of HPV-16 infected women are seroconverted between 6 and 18 months after HPV DNA has been detected and that this rarely occurs in patients detected as having transient HPV DNA.

However, other serological studies have shown that 20-50% of women suffering from HPV-associated lesions, with HPV DNA presence, do not present detectable levels of anti-VLP antibodies; this is in part due to the lack of an optimized test and the fact that these antibodies reactivity is type-specific for the virus. An optimized VLP-based ELISA test has been recently reported showing 93% sensitivity and 98.5% specificity for discriminating between positive and negative control sera. However, there was no report to evaluate the antibody response in patients with HPV-infected cervical lesions and with the prognosis of these patients.

So in the present proposal, we would like to examine the anti-L1 antibodies of various HPV types among Taiwanese women with HPV-related CIN or cervical cancer. The purposes of this proposal are 1) to address the immunologic responses to HPV between CIN and cervical cancer patients. , 2) to elucidate the correlation between immunologic responses to HPV and disease severity of cervical cancer., 3) to evaluate the correlation between immunologic responses to HPV and the prognosis of cervical cancer patients.

The samples of patients' sera were collected on the day of surgery. 2. The sera samples were freezedon -200C until analyzed. 3. The sera samples will be shipped to the Lab. of Merck company in US. 4. HPV Serologic Assay A competitive radioimmunoassay developed by Merck Research Laboratories will be was used and perform to quantitate serum HPV- 6, 11, 16, 18, 31, 33, 45, 51, 52, 58, 59, or 68 antibodies in Merck Research Laboratories (12). Results will be read from a standard curve, corrected for dilution, and reported in arbitrary units (milli-Merck Units, or mMU per milliliter). A fixed cutoff of 5.9 mMU per milliliter (derived by repeatedly testing a panel of positive and negative samples against the standard curve) will be used to determine the HPV-6, 11, 16, 18, 31, 33, 45, 51, 52, 58, 59, or 68 serologic status of the women.

ELIGIBILITY:
Inclusion Criteria:

1. cervical intrapeithelial neoplasm
2. Cervical cancer

Exclusion Criteria:

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2005-12; Primary Completion 2006-01 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | from CS operation to close

CONTACTS AND LOCATIONS:
Overall Officials: Chi-An Chen, MD, Study Chair — National Taiwan University Hospital; Chi-An Chen, MD, Study Chair — National Taiwan Univ. Hosp.
Locations (1):
- Natioanal Taiwan Univ. Hospital, Taipei, Taiwan, China